CLINICAL TRIAL: NCT06060847
Title: Liver Resection and Simultaneous Sleeve Gastrectomy for HCC Related to Metabolic Syndrome (LIRESS)
Brief Title: Liver Resection and Simultaneous Sleeve Gastrectomy for MS-HCC (LIRESS)
Acronym: LIRESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale V. Fazzi (Other)
Responsible Party: Principal Investigator, Annarita Libia, Doctor, Ospedale V. Fazzi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/2023
Record Dates: First submitted 2023-09-08; First posted 2023-09-29 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma, Hepatocellular; Metabolic Syndrome
Keywords: hepatocellular carcinoma; sleeve gastrectomy; morbid obesity
MeSH Terms: conditions — Carcinoma, Hepatocellular; Metabolic Syndrome; Obesity, Morbid | interventions — Hepatectomy

STUDY DESIGN:
Intervention Model Description: Patients 18 years old and older, affected by hepatocellular carcinoma (HCC) with metabolic syndrome (MS) as unique risk factor, with compensated liver function (Child A) who are deemed suitable for liver resection and comply with the criteria for bariatric surgery, will undergo liver resection of HCC and simultaneous sleeve gastrectomy for morbid obesity during the same surgical procedure.
  Patients affected by HCC related to metabolic syndrome who fall within exclusion criteria, will undergo liver resection for HCC without sleeve gastrectomy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients affected by HCC induced by metabolic syndrome as unique risk factor (Experimental): Patients aged 18 years old and older, affected by HCC with MS (metabolic syndrome) as unique risk factor who comply with the criteria for bariatric surgery, will undergo liver resection and sleeve gastrectomy with minimally-invasive technique in the same surgical procedure
  Interventions: Procedure: Liver resection and simultaneous sleeve gastrectomy for HCC induced by metabolic syndrome
- Patients with HCC related to metabolic syndrome as unique risk factor (Active Comparator): Patients aged 18 years old and older, affected by HCC (hepatocellular carcinoma) with MS (metabolic syndrome) as unique risk factor who will undergo liver resection only
  Interventions: Procedure: Liver resection for HCC induced by metabolic syndrome

INTERVENTIONS:
Procedure: Liver resection and simultaneous sleeve gastrectomy for HCC induced by metabolic syndrome — Patients in the experimental arm will undergo liver resection for HCC and sleeve gastrectomy for MS during the same surgical procedure.
  Arms: Patients affected by HCC induced by metabolic syndrome as unique risk factor
Procedure: Liver resection for HCC induced by metabolic syndrome — Patients in the active comparator arm will undergo liver resection for HCC
  Arms: Patients with HCC related to metabolic syndrome as unique risk factor

SUMMARY:
Hepatocellular carcinoma (HCC) related to metabolic syndrome (MS) as unique risk factor is gradually overpassing the more common viral and alcohol etiology, becoming a global health issue. Liver surgery for metabolic syndrome-related HCC in this frail subset of patients constitute a challenge, due to high morbidity and mortality rate reported in literature, and contrasting results in term of oncologic outcome. The present multicentric prospective study aims to ascertain if the combination of sleeve gastrectomy and liver surgery in the same surgical procedure may have benefit in terms of reduced perioperative morbidity and prolonged Overall Survival and Recurrence Free Survival. Secondary outcome will be the evaluation of the consequences induced by sleeve gastrectomy on liver disease, in particular liver fibrosis evaluated in term of NFS score (Non-Alcoholic Fatty Liver Disease Fibrosis score), FIB-4 (Fibrosis-4 Index for Liver Fibrosis) score and Fibroscan transient elastography.

DETAILED DESCRIPTION:
Obesity is a worldwide epidemic, with more than 2 billion people currently overweight and an additional 1.12 billion projected to be overweight by 2030. HCC (hepatocellular carcinoma) associated to obesity and its comorbidity is overcoming Hepatitis C Virus (HCV) related cancer and is already the leading cause of liver transplant in USA. HCC remains the sixth most common cancer in the world and the third cause of cancer-related death. Considering these epidemiological evidence, the incidence of MS-HCC (metabolic syndrome-related hepatocellular carcinoma) is expected to increase with huge cost efforts for the global healthcare system. The impaired performance status of patients with HCC and metabolic syndrome seems to explain high perioperative morbidity rate reported in literature. Literature reports several experiences of bariatric surgery combined to liver transplant for chronic liver disease related induced by non alcoholic steatohepatitis (NASH), performed before or after liver surgery, or even at the same time. Even if evidences are weak, outcomes reported seem to be promising. Since sleeve gastrectomy is not only a mere restrictive bariatric procedure, but it produces hormonal and metabolic changes, with the present study the investigators want to ascertain if sleeve gastrectomy at time of liver resection for MS-HCC (metabolic syndrome-related hepatocellular carcinoma) can modify short perioperative outcomes and long-term oncologic results.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial
2. Be ≥ 18 years of age on day of signing informed consent.
3. Have hepatocellular carcinoma with metabolic syndrome as unique risk factor
4. Have an overall Child-Pugh score = A
5. Be eligible for liver resection with laparoscopic or robotic technique
6. Be eligible for bariatric surgery as defined below

   * BMI ≥ 40 kg/m2
   * BMI ≥ 35-40 kg/m2 with associated comorbidities
   * BMI 30-35 kg/m2 and type 2 diabetes
   * BMI 30-35 kg/m2 and arterial hypertension with poor control despite optimal medical therapy.

Exclusion Criteria:

1. Have hepatocellular carcinoma related to other etiology, even in case of coexisting metabolic syndrome
2. Denial of the patient to undergo bariatric procedure
3. Have BMI < 30
4. Have negative opinion of psychologic consultant
5. Have an overall Child-Pugh score > 7
6. Evidence of clinical significant portal hypertension as followed:

   * esophageal varices
   * gastric varices
   * portal hypertensive gastropathy
   * gastric vascular ectasia

Of note: 1) Conversion to open surgery for any reason does not represent a reason of data exclusion from the analysis; 2) any type of hepatic resection, according to Brisbane classification, is included, also major hepatectomy requiring preoperative intervention to achieve adequate volume remnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-06 (Estimated); Primary Completion 2029-03-06 (Estimated); Study Completion 2032-03-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 year, 3 years, 5 years
  Calculated from the date of diagnosis to the date of death from any cause
Recurrence-free Survival | 1 year, 3 years, 5 years
  Calculated from the date of surgery to the date of recurrence
90-day mortality | 90 post-operative days
  Mortality from any cause
Comprehensive Complication Index | 90 post-operative days
  Any deviation from the normal postoperative course measured on a scale from 0 (no complication) to 100 (death)

SECONDARY OUTCOMES:
Fibrosis-4 Index for Liver Fibrosis score | After 6 months, up to 5 years
  Fibrosis-4 Index for Liver Fibrosis score (FIB-4 score) will be calculated using the following formula:
  FIB-4 score= Age (years)× aspartate aminotransferase (AST) (U/L)/[platelet count (109/L)×√alanine aminotransferase (ALT) (U/L)]
Non-Alcoholic Fatty Liver Disease Fibrosis Score | After 6 months, up to 5 years
  Non-Alcoholic Fatty Liver Disease Fibrosis Score (NFS score) will be calculated using the following formula:
  NFS = -1.675 + 0.037 - age (years) + 0.094 - BMI (kg/m2) + 1.13 × impaired fasting glucose/diabetes (yes = 1, no = 0) + 0.99 × aspartate aminotransferase/ alanine aminotransferase (AST/ALT) ratio - 0.013 × platelet count (×109/l) - 0.66 × albumin (g/dl).
Fibroscan stiffness | After 6 months, up to 5 years
  The Fibroscan stiffness measurement relies on the propagation of elastic waves to assess the stiffness of the liver: the faster elastic waves propagates within the liver, the stiffer the organ is. The final liver stiffness value is the median of individual liver stiffness values using the valid measurements and is expressed in kilo Pascal (kPa).
Body Mass Index | After 3 months, up to 5 years
  Body Mass Index (BMI) is combination of bodyweight and body height and presented as kg/m^2
Weight loss | After 3 months, up to 5 years
  Weight loss expressed in Kg
Percent excess weight loss | After 3 months, up to 5 years
  Percent excess weight loss (%EWL) is calculated as follows: [(initial weight - current weight) / (initial weight - ideal weight)] × 100
Control of obesity-induced hypertension | After 3 months, up to 5 years
  Change of antihypertensive therapy assessed by medical history questionnaire
Control of obesity-induced comorbidities | After 3 months, up to 5 years
  change of insulin therapy or oral hypoglycemics assessed by medical history questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Annarita Libia, Principal Investigator — Ospedale Vito Fazzi, Lecce
Locations (1):
- Ospedale Vito Fazzi, Lecce, Italy

REFERENCES:
- [Background] Yang T, Hu LY, Li ZL, Liu K, Wu H, Xing H, Lau WY, Pawlik TM, Zeng YY, Zhou YH, Gu WM, Wang H, Chen TH, Han J, Li C, Wang MD, Wu MC, Shen F. Liver Resection for Hepatocellular Carcinoma in Non-alcoholic Fatty Liver Disease: a Multicenter Propensity Matching Analysis with HBV-HCC. J Gastrointest Surg. 2020 Feb;24(2):320-329. doi: 10.1007/s11605-018-04071-2. Epub 2019 Jan 7. PMID 30617773
- [Background] Cauchy F, Zalinski S, Dokmak S, Fuks D, Farges O, Castera L, Paradis V, Belghiti J. Surgical treatment of hepatocellular carcinoma associated with the metabolic syndrome. Br J Surg. 2013 Jan;100(1):113-21. doi: 10.1002/bjs.8963. Epub 2012 Nov 12. PMID 23147992
- [Background] de Barros F, Cardoso Faleiro Uba PH. Liver transplantation and bariatric surgery: a new surgical reality: a systematic review of the best time for bariatric surgery. Updates Surg. 2021 Oct;73(5):1615-1622. doi: 10.1007/s13304-021-01106-3. Epub 2021 Jun 12. PMID 34118015
- [Background] Hobeika C, Ronot M, Beaufrere A, Paradis V, Soubrane O, Cauchy F. Metabolic syndrome and hepatic surgery. J Visc Surg. 2020 Jun;157(3):231-238. doi: 10.1016/j.jviscsurg.2019.11.004. Epub 2019 Dec 19. PMID 31866269